CLINICAL TRIAL: NCT03810911
Title: Mechanisms of Erythropoietin Induced Hypertension
Brief Title: Mechanisms of EPO-induced Hypertension
Acronym: EPIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped because of inability to reach target sample size.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEPH-005-18S; 052387 (Other Grant/Funding Number: Indiana Institute for Medical Research)
Record Dates: First submitted 2019-01-07; First posted 2019-01-22 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease; Blood Pressure; Anemia
Keywords: Flow mediated dilatation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: All subjects will receive darbepoetin during the study. One group, the immediate start group, will receive the drug the day of randomization. The other group, the delayed start group, will receive the drug 12 weeks later.
Masking Description: The groups are randomized not the study drug. The groups will be known by both the participant and the investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early start (Active Comparator): Participants given study drug immediately at randomization
  Interventions: Drug: Darbepoetin
- Delayed start (No Intervention): Participants given study drugs 12 weeks after randomization

INTERVENTIONS:
Drug: Darbepoetin — Used to treat anemia. In the group labeled no intervention, the intervention is simply delayed 12 weeks after randomization as noted in the description.
  Other Names: EPO
  Arms: Early start

SUMMARY:
The investigators hypothesize that compared to untreated controls, erythropoietin (EPO) therapy in anemic patients with chronic kidney disease will raise diastolic blood pressure (BP). The magnitude of increase in diastolic BP at 12 weeks after treatment will be related to two factors. First, endothelial dysfunction and worsening of endothelial function from baseline to 4 weeks and second, the change of forearm blood flow in response to breathing oxygen and the change in this measure from baseline to 4 weeks. Study procedures include fasting blood draws, ambulatory blood pressure, urine collection, and forearm blood flow tests. The study hopes to accrue 160 subjects.

DETAILED DESCRIPTION:
Hypertension is a common but frequently overlooked and underreported adverse effect of erythropoietin (EPO) therapy. Recent trials have noted substantial cardiovascular risks associated with normalization of hemoglobin. The risk of strokes is strongly related to poorly controlled hypertension. Blood pressure was not measured the way it usually is in hypertension trials, so the investigators cannot be completely confident that the risk of strokes in this large randomized trial was not related to EPO-induced hypertension. New therapies, such as hypoxia-inducible factor (HIF) stabilizers are on the horizon but it remains to be seen whether these new drugs would have a lower or a higher risk for hypertension compared to EPO. Accordingly, understanding the mechanism of EPO-induced hypertension is urgent. The investigators hypothesize that compared to untreated controls, EPO therapy in anemic patients with chronic kidney disease (CKD) will raise diastolic blood pressure. The magnitude of increase in diastolic BP at 12 weeks after treatment will be related to endothelial dysfunction and worsening of endothelial function from baseline to 4 weeks. If the investigators understood the time course, the magnitude, and the mechanisms of EPO-induced hypertension (EIH) the investigators will better be able to design studies to compare the vascular effects of EPO and HIF stabilizers in the future. Thus, this study has the potential of improving the investigators' understanding of a common side effect of EPO by precisely quantifying the magnitude of BP change, its effects on endothelial function, and discovering the biomarkers of these adverse effects. Thus, the investigators can in the future robustly compare these effects of EPO with HIF stabilizers. This study is innovative because it will focus on the potential mechanisms by which EPO induces an increase in BP. The time-course and magnitude of change in BP will be assessed using the gold-standard measurement of 24 hour ambulatory BP recordings. The more frequent clinic BP recordings using validated methods will better allow us to track changes in BP over time. The investigators' lab is uniquely qualified to carry out these experiments due to a large experience with such types of studies. The investigators will examine endothelial function using a reference method -- that of flow-mediated dilatation -- which is established in the investigators' laboratory. The investigators will directly test the hypothesis whether endothelial function is responsible for the BP increase.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3 or 4 chronic kidney disease
* Controlled hypertension with 24 hour ambulatory blood pressure monitoring less than 140/90 mmHg at baseline and treatment with at least 1 antihypertensive medication
* Hemoglobin between 8 and 10 g/dL
* No treatment with erythropoiesis-stimulating agents (ESA) within 3 previous months

Exclusion Criteria:

* Need for packed red blood cells (RBC) transfusion in the previous 2 months
* Myocardial infarction, stroke or hospitalization for heart failure in the past 2 months
* In the assessment of the investigator, have hematologic, inflammatory, infectious, or other conditions that might interfere with the erythropoietic response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD MBBS, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Georgianos PI, Agarwal R. Resistant Hypertension in Dialysis: Epidemiology, Diagnosis, and Management. J Am Soc Nephrol. 2024 Apr 1;35(4):505-514. doi: 10.1681/ASN.0000000000000315. Epub 2024 Jan 16. PMID 38227447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 18 December 2020, and 22 September 2023, 1699 individuals were assessed for study eligibility. These individuals were screened, 4398 times for a mean of 2.6 times per person. In all, 281 (17%) were noted to be potentially eligible, of which, 157 (56%) agreed to come for a consent visit.
Pre-assignment Details: 65 individuals (41%) consented, of which, 27 (42%) were enrolled in the trial and underwent randomization stratified by the level of albuminuria (KDIGO stage A1, A2, or A3). 16 were assigned to waitlisted and 11 to immediate start group. In each of the two groups, two patients did not complete the study. The most common reason for randomization failure was either Hgb out of range (39%) or ambulatory BP out of range (39%). The trial was stopped because of inability to reach target sample size.
Period: Overall Study
Arm/Group | Early Start | Delayed Start
Started | 11 | 16
Completed | 9 | 14
Not Completed | 2 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomization was stratified by the level of albuminuria in a 1:1 ratio to either early or delayed treatment with ESA. A random permuted block design was used to avoid imbalance in assignment to the study drugs over time. After confirming eligibility, the principal investigator used a computer program to reveal the group assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Start | Delayed Start | Total
Number analyzed (Participants) | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self stated race: White | 10 | 9 | 19
  Self stated race: Black | 1 | 7 | 8
Weight -- kg (SD) [Mean (Standard Deviation); unit: kg] | 99.3 (19.7) | 88.5 (24.5) | 92.9 (22.9)
Age, Customized [Mean (Standard Deviation); unit: Years]
  Age - years (SD) | 74.6 (6) | 75.1 (9.3) | 74.9 (8)
Medical History [Count of Participants; unit: Participants]
  Diabetes -- n (%) | 8 | 9 | 17
  Myocardial infarction -- n (%) | 2 | 4 | 6
  Stroke -- n (%) | 1 | 1 | 2
  Coronary revascularization -- n (%) | 4 | 6 | 10
  Heart failure hospitalization -- n (%) | 5 | 5 | 10
Hemoglobin -- g/dL (SD) [Mean (Standard Deviation); unit: g/dL] | 9.4 (0.6) | 9.5 (0.7) | 9.4 (0.6)
Serum ferritin -- ng/mL (25th-75th percentile) [Mean (Inter-Quartile Range); unit: ng/mL] | 110 [11 to 194] | 91 [40 to 434] | 95 [38 to 353]
Transferrin saturation -- percent (SD) [Mean (Standard Deviation); unit: %] | 21 (9.8) | 24.2 (15.5) | 23 (13.3)
Baseline eGFR -- mL/min/1.73m^2 (SD) [Mean (Standard Deviation); unit: mL/min/1.73m^2] — Estimated glomerular filtration rate (eGFR) is an estimate of kidneys' ability to filter blood. A lower eGFR can indicate a greater risk or progression of CKD. An eGFR <60 ml/min/1.73 m² that persists for a minimum of 3 months indicates the presence of CKD.
  mL/min/1.73m^2 | 38.6 (11.7) | 36 (13.9) | 37.1 (12.9)
Glomerular filtration rate (GFR) category (G1-G5) [Count of Participants; unit: Participants] — KDIGO glomerular filtration rate (GFR) category (G1-G5) is one marker of CKD. The categories are defined as the following and must be present for at least 3 months (ml/min/1.73):
  G1 - GFR range: ≥ 90 G2 - GFR range: 60-89 G3a - GFR range: 45-59 G3b - GFR range: 30-44 G4 - GFR range: 15-29 G5 - GFR range: < 15 A lower eGFR, or a higher eGFR category, can indicate a greater progression or risk of CKD. This study included only patients with Stage 3 or 4 CKD defined as eGFR category G3 or G4 or those with persistent albuminuria category A2 or A3, hence the single participant in G2.
  Participants
    G2 -- n (%) | 0 | 1 | 1
    G3a -- n (%) | 5 | 3 | 8
    G3b -- n (%) | 4 | 6 | 10
    G4 -- n (%) | 2 | 6 | 8
Albuminuria category (A1-A3) [Count of Participants; unit: Participants] — KDIGO persistent albuminuria category is one marker of CKD. The categories are defined as the following using urine-albumin-to-creatinine ratio (UACR) and must be present for at least 3 months (mg/g):
  A1 - UACR range: <30 A2 - UACR range: 30-300 A3 - UACR range: >300 A greater the amount of albuminuria, or a higher persistent albuminuria category, can indicate a greater progression or risk of CKD. This study included only patients with Stage 3 or 4 CKD defined as eGFR category G3 or G4 or those with persistent albuminuria category A2 or A3, hence the single participant in G2.
  Participants
    A1 -- n (%) | 4 | 5 | 9
    A2 -- n (%) | 5 | 8 | 13
    A3 -- n (%) | 2 | 3 | 5
Baseline UACR -- mg/g creatinine median (25th-75th) [Median (Inter-Quartile Range); unit: mg/g] — Urine albumin-to-creatinine ratio (UACR) is a measurement of the amount of protein (albumin) in a patient's urine. A UACR ≥30 mg/g indicates the presence of albuminuria, and greater UACR value can indicate a greater risk or progression of CKD.. A UACR ≥30 mg that persists for a minimum of 3 months indicates the presence of CKD.
  mg/g | 39 [15 to 60] | 79 [16 to 191] | 56 [15 to 183]
Baseline clinic blood pressure [Mean (Standard Deviation); unit: mmHg]
  Clinic systolic blood pressure -- mmHg (SD) | 125.1 (22.1) | 123.2 (15.8) | 124.4 (19.5)
  Clinic diastolic blood pressure -- mmHg (SD) | 58.5 (12.1) | 55.4 (10.6) | 57.2 (11.4)
Antihypertensive drugs -- n (SD) [Mean (Standard Deviation); unit: Drugs] | 3.5 (1.2) | 3 (1.2) | 3.2 (1.2)
Nature of antihypertensive drugs [Count of Participants; unit: Participants]
  ACE inhibitors or ARBs -- n (%) | 7 | 6 | 13
  K sparing diuretics -- n (%) | 2 | 3 | 5
  Loop diuretics -- n (%) | 5 | 4 | 9
  Thiazide diuretics -- n (%) | 4 | 4 | 8
  Dihydropyridine Ca channel blockers -- n (%) | 6 | 9 | 15
  Nondihydropyridine Ca channel blockers -- n (%) | 1 | 0 | 1
  Beta blockers -- n (%) | 7 | 14 | 21
  Alpha blockers -- n (%) | 5 | 3 | 8
  Vasodilators -- n (%) | 1 | 5 | 6
Clinic heart rate -- beats per minute (SD) [Mean (Standard Deviation); unit: beats per minutes] | 71 (8) | 65 (10) | 68 (9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Diastolic Blood Pressure in EPO Treated Patients Compared to Delayed Start Controls
Description: In the delayed start group (the control group), the investigators will measure the change in diastolic blood pressure from 0 weeks to 12 weeks compared to the change in diastolic BP from 0 to 12 weeks in the immediate start group.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Early Start | Delayed Start
Number analyzed (Participants) | 11 | 16
mmHg | 1.4 [-1.8 to 4.6] | -0.5 [-4.7 to 3.8]

2. Secondary Outcome: Change in Systolic Blood Pressure in EPO Treated Patients Compared to Delayed Start Controls
Description: In the delayed start group (the control group), the investigators will measure the change in systolic blood pressure change from 0 weeks to 12 weeks compared to the change in systolic BP from 0 to 12 weeks in the immediate start group.
Time Frame: Baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Early Start | Delayed Start
Number analyzed (Participants) | 11 | 16
mmHg | 2 [-3.9 to 7.9] | -3.6 [-11.5 to 4.3]

3. Secondary Outcome: Number of Participants With Worsened Hypertension Status in Immediate Start Group Compared to Delayed Start Controls
Description: Worsening of hypertension at any time point will be defined as either an increase in blood pressure medication, an increase in seated clinic diastolic blood pressure by greater than or equal to 10 mmHg or systolic blood pressure increase of greater than or equal to 20 mmHg. Between-group change in hypertension status from baseline to 12 weeks will be compared in the immediate start and delayed start groups.
Time Frame: Baseline to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Early Start | Delayed Start
Number analyzed (Participants) | 11 | 16
Participants | 3 | 7

4. Secondary Outcome: Number of Participants With Worsened Hypertension Status in Delayed Start Group Participants When They Were Not on EPO Compared to When They Were on EPO
Description: Worsening of hypertension at any time point will be defined as either an increase in blood pressure medication, an increase in seated clinic diastolic blood pressure by greater than or equal to 10 mmHg or systolic blood pressure increase of greater than or equal to 20 mmHg. Within-group change in hypertension status from 12 weeks to 24 weeks will be compared to the control period of 0 weeks to 12 weeks in the delayed start group.
Time Frame: baseline to 12 weeks vs 12 weeks to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- No Darbepoetin: Data collected from the delayed start group from baseline to 12 weeks when participants were not taking darbepoetin
- Darbepoetin: Data collected from the delayed start group from 12 weeks to 24 weeks when participants were taking darbepoetin
Arm/Group | No Darbepoetin | Darbepoetin
Number analyzed (Participants) | 16 | 16
Participants | 7 | 7

5. Secondary Outcome: Change in Endothelial Function in Those Treated With EPO Compared to the Waitlisted Group
Description: The investigators used the high-resolution ultrasound of brachial artery to assess flow-mediated dilatation (FMD). FMD measures the dilation of blood vessels in response to increased blood flow and is the reference standard for assessing endothelial function. The mean percentage change in endothelial function of those treated with EPO were compared to that of the delayed start group. The hypothesis being tested is that EPO will cause impairment in endothelial function.
Time Frame: Baseline to 4 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of endothelial function
Arm/Group | Early Start | Delayed Start
Number analyzed (Participants) | 11 | 16
percentage of endothelial function | 0.9 [-3 to 4.8] | -1.2 [-4 to 1.6]

6. Primary Outcome: Within Group Change in Diastolic Blood Pressure in the Delayed Start Group
Description: Within group change in diastolic blood pressure from 12 weeks to 24 weeks compared to change in diastolic blood pressure from baseline to 12 weeks in the delayed start group
Time Frame: 12 to 24 weeks compared to baseline to 12 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | No Darbepoetin | Darbepoetin
Number analyzed (Participants) | 16 | 14
mmHg | -1.9 [-5.4 to 1.6] | 3.2 [-0.5 to 6.8]

7. Secondary Outcome: Change in Urine Albumin to Urine Creatinine Ratio in the Delayed Start Group
Description: Change in urine albumin to urine creatinine ratio in the delayed start group baseline to 16 weeks (which is 4 weeks of exposure to darbepoetin), from baseline to 20 weeks (8-week exposure), and from baseline to 24 weeks (12-week exposure)
Time Frame: Baseline to 16 weeks, baseline to 20 weeks, and baseline to 24 weeks
Measure: Mean (95% Confidence Interval); unit: percentage change in UACR from baseline
Groups:
- 16 Weeks (4-week Darbepoetin Exposure): Data from the delayed start group baseline to 16 weeks (4-week darbepoetin exposure)
- 20 Weeks (8-week Darbepoetin Exposure): Data from delayed start group baseline to 20 weeks (8-week darbepoetin exposure)
- 24 Weeks (12-week Darbepoetin Exposure): Data from delayed start group baseline to 24 weeks (12-week darbepoetin exposure)
Arm/Group | 16 Weeks (4-week Darbepoetin Exposure) | 20 Weeks (8-week Darbepoetin Exposure) | 24 Weeks (12-week Darbepoetin Exposure)
Number analyzed (Participants) | 16 | 16 | 16
percentage change in UACR from baseline | 22 [0 to 65] | 22 [0 to 49] | 35 [11 to 82]

ADVERSE EVENTS:
Time Frame: through study completion, at most 6 months
Description: Harms will be assessed by monitoring changes in weight, eGFR, CBC, clinic BP, and ABPM. Safety of continued participation will be assessed at each study visit. The stop-points will be treatment-emergent severe adverse events that precludes further exposure to the drug, such as an allergic drug reaction, initiation of renal replacement therapy, or death. If the study drug is stopped, the subject will be continued to be studied so as to not violate the intention-to-treat principle.
Groups:
- Darbepoetin: Data from participants that were actively taking darbepoetin at the time of collection
- No Darbepoetin: Data from participants that were not taking darbepoetin at the time of collection
Arm/Group | Darbepoetin | No Darbepoetin
All-Cause Mortality (participants affected / at risk) | 2/27 | 0/16
Serious Adverse Events (participants affected / at risk) | 8/27 | 5/16
Other Adverse Events (participants affected / at risk) | 6/27 | 7/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin (N=27) | No Darbepoetin (N=16)
Falls (General disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 3 (4) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Hypertensive crisis (Cardiac disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Cardiac disorders) | 1 (1) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Venous thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Abnormal renal labs (Renal and urinary disorders) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right leg weakness following cardiac catheterization (General disorders) | 0 (0) | 1 (1)
Unfit living conditions (General disorders) | 1 (1) | 0 (0)
Acute cholecystitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin (N=27) | No Darbepoetin (N=16)
Falls (General disorders) | 0 (0) | 1 (2)
Skin irritation or rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypoglycemia (General disorders) | 1 (1) | 0 (0)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Delerium (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Kidney transplant hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was limited by the absence of enough patients to observe a meaningful change in 24-hour ambulatory BP or endothelial function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03810911/Prot_SAP_000.pdf